CLINICAL TRIAL: NCT06078475
Title: Efficacy Of Modified Perichondral Approach Thoracoabdominal Nerve Block For Post Cesarean Section Pain
Brief Title: Efficacy of Modified Perichondral Approach Thoracoabdominal Nerve Block For Post Cesarean Section
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa City Hospital (Other Government)
Responsible Party: Principal Investigator, Mursel Ekinci, assoc prof, Bursa City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Bursa City Hospital 3
Record Dates: First submitted 2023-07-25; First posted 2023-10-11 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Cesarean Section
Keywords: Cesarean Section Pain; Postoperative Analgesia; Modified Perichondral Approach Thoracoabdominal Nerve Block

STUDY DESIGN:
Intervention Model Description: There are two models for this study. Modified Perichondral Approach Thoracoabdominal Nerve block (M-TAPA block) group, and Control (C) group
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient and the outcomes assessor who performs postoperative pain evaluation will not know the group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group M-TAPA (Modified Perichondral Approach Thoracoabdominal Nerve block group) (Active Comparator): In group M-TAPA, M-TAPA block will be performed with patient is in the supine position. After providing aseptic conditions, the high frequency linear US probe (11-12 MHz, Vivid Q) will be covered with a sterile sheath, and an 80 mm block needle (Braun 360°) will be used. The US probe will be placed in the sagittal plane where the midclavicular line intersects with the costal cartilage corresponding to the costochondral angle. Using the In Plane technique, the probe is gently pushed to visualize the lower part of the costochondral angle at the central level, advancing the block needle in the caudal-cranio direction, 5 ml of saline will be injected into the layer between the transverse abdominal muscle and the lower plane of the costal cartilage, and the block location will be confirmed. After the block location is confirmed, a total of 20 ml + 20 ml of 0.25% bupivacaine(Buvasin %5 flakon) (total 40 ml for both sides) will be injected bilaterally.
  Interventions: Other: Postoperative analgesia management
- Group C (Control group) (Active Comparator): In the control group, analgesics will be administered according to the protocol in postoperative analgesia management.
  Interventions: Other: Postoperative analgesia management

INTERVENTIONS:
Other: Postoperative analgesia management — Patients will be administered paracetamol 1 gr (PERFALGAN® ) IV every 8 hours in the postoperative period.. If the patient's NRS score is ≥ 4 0,5 mg/kg IV meperidine (Aldolan ampul 100 mg/2 ml) will be administered.

SUMMARY:
Cesarean section (CS) is one of the most frequently performed surgical procedures in the World. Moderate to severe postoperative pain occurs in a significant proportion of women after cesarean surgery.

Modified Perichondral Approach Thoracoabdominal Nerve (M-TAPA) block performed with ultrasound (US) is a novel technique that provides effective analgesia in the anterior and lateral thoracoabdominal areas, where local anesthetic is applied only to the lower side of the perichondral surface. M-TAPA block is a good alternative for analgesia of the upper dermatome levels and the abdominal lateral Wall, provides analgesia in the abdominal area at the T5-T11 level.

The aim of this study is to evaluate the effectiveness of US-guided M-TAPA block for postoperative analgesia management after cesarean section.

DETAILED DESCRIPTION:
Cesarean section (CS) is one of the most frequently performed surgical procedures in the World, in European countries, approximately 20% of deliveries are CS. Moderate to severe postoperative pain occurs in a significant proportion of women after cesarean surgery. This delays recovery and returning to daily life. Postoperative pain disrupts the mother-child bond, makes breastfeeding difficult, and affects the psychological state of the mother. Also inadequate postoperative analgesia may cause hyperalgesia and chronic pain.

Perioperative pain should be managed with a multi-modal approach. Opioids and nonsteroid anti inflammatory drugs should be considered as components of a multimodal analgesic regimen. However, use of both systemic and neuraxial opioids may be associated with effects (respiratory depression, nausea, vomiting, sedation, pruritus, hyperalgesia). For this, interfacial blocks may be preffered to provide postoperative analgesia and reduced opioid consumption.

Modified Perichondral Approach Thoracoabdominal Nerve (M-TAPA) block performed with ultrasound (US) is a novel technique that provides effective analgesia in the anterior and lateral thoracoabdominal areas, where local anesthetic is applied only to the lower side of the perichondral surface. M-TAPA block is a good alternative for analgesia of the upper dermatome levels and the abdominal lateral Wall, provides analgesia in the abdominal area at the T5-T11 level. Sonoanatomy is easy to visualize and the spread of local anesthetic can be easily seen under US guidance.

In the literature, there are studies investigating the effectiveness of M-TAPA block for post-operative pain management in bariatric surgery. However, there is no randomized study evaluating the effectiveness of M-TAPA block for postoperative analgesia management after CS. The aim of this study is to evaluate the effectiveness of US-guided M-TAPA block for postoperative analgesia management after cesarean section. The primary outcome is to compare global recovery scores, the secondary outcome is to compare postoperative pain scores (NRS), to evaluate postoperative rescue analgesic (opioid) use and side effects (allergic reaction, nausea, vomiting) associated with opioid use in this study.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) classification II
* Elective cesarean section, and gestational age above 37 weeks will be included

Exclusion Criteria:

* Bleeding diathesis
* Anticoagulant treatment
* Local anesthetics and opioid allergy
* Infection at the site of block
* Patients who do not accept the procedure

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-05-15 (Estimated)

PRIMARY OUTCOMES:
Global recovery scoring system (patient satisfaction scale) | The quality of recovery will be evaluated out of a total of 150 points according to the QoR-15 test to be applied at the portoperative 24th hour.
  We will use the Turkish version of Quality of Recovery / QoR-15 questionairre
  PART A How have you been feeling in the last 24 hours? (0 to 10, where: 0 = none of the time [poor] and 10 = all of the time [excellent])
  1. Able to breathe easily
  2. Been able to enjoy food
  3. Feeling rested
  4. Have had a good sleep
  5. Able to look after personal toilet and hygiene unaided
  6. Able to communicate with
  7. Getting support from hospital doctors and nurses
  8. Able to return to work or usual home activities
  9. Feeling comfortable and in control
  10. Having a feeling of general well-being
      PART B Have you had any of the following in the last 24 hours? (10 to 0, where: 10 = none of the time [excellent] and 0 = all of the time [poor])
  11. Moderate pain
  12. Severe pain
  13. Nausea or vomiting
  14. Feeling worried or anxious
  15. Feeling sad or depressed

SECONDARY OUTCOMES:
Postoperative pain scores (Numerical rating scale) (0-meaning "no pain" to 10-meaning "worst pain imaginable") | Patients will be evaluated at the first 24 hours period postoperatively.
  Postoperative 24 hours period. Patients' pain scores will be questioned at 0, 2, 4, 8, 16 and 24 hours.
The use of rescue analgesia | Meperidine consumption will be recorded at the first 24 hours period postoperatively. (Number of Participants and Concentration of Meperidin)
  The need for rescue analgesia will be recorded at the first 24 hours period postoperatively.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - T.C. Sağlık Bakanlığı Bursa Şehir Hastanesi, Bursa
  - Mursel Ekinci, Bursa

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared

REFERENCES:
- [Background] Riemma G, Schiattarella A, Cianci S, La Verde M, Morlando M, Sisti G, Esposito I, Della Corte L, Sansone P, De Franciscis P. Transversus abdominis plane block versus wound infiltration for post-cesarean section analgesia: A systematic review and meta-analysis of randomized controlled trials. Int J Gynaecol Obstet. 2021 Jun;153(3):383-392. doi: 10.1002/ijgo.13563. Epub 2021 Feb 11. PMID 33368204
- [Background] Kintu A, Abdulla S, Lubikire A, Nabukenya MT, Igaga E, Bulamba F, Semakula D, Olufolabi AJ. Postoperative pain after cesarean section: assessment and management in a tertiary hospital in a low-income country. BMC Health Serv Res. 2019 Jan 25;19(1):68. doi: 10.1186/s12913-019-3911-x. PMID 30683083
- [Background] Kara U, Simsek F, Kamburoglu H, Ozhan MO, Alakus U, Ince ME, Eksert S, Ozkan G, Eskin MB, Senkal S. Linguistic validation of a widely used recovery score: quality of recovery-15 (QoR-15). Turk J Med Sci. 2022 Apr;52(2):427-435. doi: 10.55730/1300-0144.5330. Epub 2022 Apr 14. PMID 36161615
- [Background] Ohgoshi Y, Ando A, Kawamata N, Kubo EN. Continuous modified thoracoabdominal nerves block through perichondrial approach (M-TAPA) for major abdominal surgery. J Clin Anesth. 2020 Mar;60:45-46. doi: 10.1016/j.jclinane.2019.08.031. Epub 2019 Aug 20. No abstract available. PMID 31442859
- [Background] Tulgar S, Selvi O, Thomas DT, Deveci U, Ozer Z. Modified thoracoabdominal nerves block through perichondrial approach (M-TAPA) provides effective analgesia in abdominal surgery and is a choice for opioid sparing anesthesia. J Clin Anesth. 2019 Aug;55:109. doi: 10.1016/j.jclinane.2019.01.003. Epub 2019 Jan 9. No abstract available. PMID 30639940